CLINICAL TRIAL: NCT03834415
Title: Influence of Lactobacillus Reuteri DSM17938 on Early Gut Microbial Colonization in Infants Born by Caesarean Section: A Double-blinded, Randomized, Placebo-controlled Study
Brief Title: Lactobacillus Reuteri DSM17938 in C-Section Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovacion y Desarrollo de Estrategias en Salud (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Pedro Gutierrez Castrellon, Head of Translational Research Center for Mother-Child Health, Innovacion y Desarrollo de Estrategias en Salud
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CSUB0153
Record Dates: First submitted 2019-02-05; First posted 2019-02-08 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-06

CONDITIONS: C-section
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: RCT two arms to evaluate the safety and efficacy of L. reuteri vs. placebo to modulate the microbiome gut profile in newborn babies delivered by C-section
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding process will be structured centrally. The oil drops of active are contained in an ambar flask. Placebo consistency, smell, flavor and container are identical to active product
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus reuteri DSM17038 (Experimental): Lactobacillus reuteri DSM17038, 1x108 CFU once a day for 30 days
  Interventions: Dietary Supplement: Lactobacillus reuteri DSM17038
- Placebo probiotics (Placebo Comparator): Placebo for probiotics, pols drops similar in consistency and flavor as experimental product
  Interventions: Other: Placebo for Probiotics

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri DSM17038 — Oil drops of L. reuteri containing 1x10>8 CFU
  Arms: Lactobacillus reuteri DSM17038
Other: Placebo for Probiotics — Oil drops mimicking in consistency and flavor to experimental product
  Arms: Placebo probiotics

SUMMARY:
RCT designed to evaluate the impact of Lactobacillus reuteri DSM17938 to modify gut microbiota in children delivered by C-section

DETAILED DESCRIPTION:
RCT designed to evaluate the safety and efficacy of L. reuteri DSM17938 administrated to newborns babies to modify the fecal microbiome after 30 days of supplementation. Secondary Secondary endpoints will be evaluate the occurrence and frequency of AEs Day 0 to Day 60; The gut bacterial composition Day 7 and Day 30 as described in primary endpoint; the gut bacterial composition in infants born by c-section and supplemented with L. reuteri DSM17938 compared to the gut bacterial composition in infants born vaginally and the salivary concentration of IgA at 48h ±3h after birth and at Day 30.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age >37weeks +0 days and <39 weeks +0 days
* Birth weight appropriate for gestational age (AGA) or Large for Gestational Age (LGA)
* Apgar score 8 or greater
* Children will receive more than 50% of the feeding occasions with human breastmilk
* Mothers will have the intention to exclusively or predominantly breastfeed the subject. On the diary report form mother will report day by day the frequency of human lactation and the frequency and amount of infant formula.
* Readiness and the opportunity for parents to fill out a study diary, questionnaires.
* Parent(s) are willing to postpone major changes in the infant feeding mode, and
* Written informed consent from parents

Exclusion Criteria:

* Older than 24 hours after birth when given the first dose of investigational product
* Any kind of chronic or acute diseases during pregnancy that can modify fecal microbiota in children, e.g. gestational diabetes, pre-clampsia, gastrointestinal disease
* Congenital malformations or anomalies
* Maternal use of antibiotics from gestational week 33 and throughout the study period.
* Maternal use of probiotics from gestational week 33 and throughout the study period.
* Maternal severe obesity at inclusion or at delivery evaluated using Rosso Madrones centiles
* Infant use of antibiotics throughout the study period.
* Infant use of probiotics throughout the study period, including infant formula and/or supplementation.
* Infants carrying out general anesthesia
* Meconium aspiration syndrome
* History of premature disruption of membranes for >24h
* Participation in other clinical trials

Ages: 12 Hours to 36 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-06-18 (Actual)

PRIMARY OUTCOMES:
Changes on fecal microbiome diversity at day 14 | 14 days
  Changes on diversity evaluated by Shannon Index of firmicutes, bacteroidetes and actinobacteria at day 14 after intervention
Changes on fecal microbiome abundance at day 14 | 14 days
  Changes on abundance evaluated by Simpson Index of firmicutes, bacteroidetes and actinobacteria at day 14 after intervention
Changes on fecal microbiome stability at day 14 | 14 days
  Changes on stability evaluated by Chao Index of firmicutes, bacteroidetes and actinobacteria at day 14 after intervention

SECONDARY OUTCOMES:
Changes on fecal microbiome diversity at day 7, 30 and 60 | 7, 30 and 60 days
  Changes on abundance evaluated by Channon Index of firmicutes, bacteroidetes and actinobacteria at day 7, 30 and 60 after intervention
Changes on fecal microbiome abundance at day 7, 30 and 60 | 7, 30 and 60 days
  Changes on abundance evaluated by Simpson Index of firmicutes, bacteroidetes and actinobacteria at day 7, 30 and 60 after intervention
Changes on fecal microbiome stability at day 7, 30 and 60 | 7, 30 and 60 days
  Changes on stability evaluated by Chao Index of firmicutes, bacteroidetes and actinobacteria at day 7, 30 and 60 after intervention
Changes on Salivary IgA levels | 7, 30 and 60 days
  Levels of salivary IgA after 7,30 and 60 days after intervention
Frequency of Adverse Event | 30 days
  Frequency of adverse events reported after randomization and until finish the treatment (day 30)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Gutierrez Castrellon, MD, MSc, DSc, Principal Investigator — Hospital General Dr. Manuel Gea Gonzalez
Locations (1):
- Hospital General Dr. Manuel Gea Gonzalez, Mexico City, Tlalpan, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Protocol documents and data base results will be available at international sites
Supporting Information: Study Protocol, SAP, CSR
Time Frame: January 2019, for 12 months
Access Criteria: IPD sharing access will be available for all investigators who want to do secondary analysis, always giving credits to principal investigators and owner of this research

REFERENCES:
- [Background] Chandel DS, Perez-Munoz ME, Yu F, Boissy R, Satpathy R, Misra PR, Sharma N, Chaudhry R, Parida S, Peterson DA, Gewolb IH, Panigrahi P. Changes in the Gut Microbiota After Early Administration of Oral Synbiotics to Young Infants in India. J Pediatr Gastroenterol Nutr. 2017 Aug;65(2):218-224. doi: 10.1097/MPG.0000000000001522. PMID 28121648
- [Background] Garcia Rodenas CL, Lepage M, Ngom-Bru C, Fotiou A, Papagaroufalis K, Berger B. Effect of Formula Containing Lactobacillus reuteri DSM 17938 on Fecal Microbiota of Infants Born by Cesarean-Section. J Pediatr Gastroenterol Nutr. 2016 Dec;63(6):681-687. doi: 10.1097/MPG.0000000000001198. PMID 27035371
- [Background] Nitert MD, Barrett HL, Foxcroft K, Tremellen A, Wilkinson S, Lingwood B, Tobin JM, McSweeney C, O'Rourke P, McIntyre HD, Callaway LK. SPRING: an RCT study of probiotics in the prevention of gestational diabetes mellitus in overweight and obese women. BMC Pregnancy Childbirth. 2013 Feb 25;13:50. doi: 10.1186/1471-2393-13-50. PMID 23442391
- [Background] Jansman AJ, Zhang J, Koopmans SJ, Dekker RA, Smidt H. Effects of a simple or a complex starter microbiota on intestinal microbiota composition in caesarean derived piglets. J Anim Sci. 2012 Dec;90 Suppl 4:433-5. doi: 10.2527/jas.53850. PMID 23365401
- [Background] Kuitunen M, Kukkonen K, Juntunen-Backman K, Korpela R, Poussa T, Tuure T, Haahtela T, Savilahti E. Probiotics prevent IgE-associated allergy until age 5 years in cesarean-delivered children but not in the total cohort. J Allergy Clin Immunol. 2009 Feb;123(2):335-41. doi: 10.1016/j.jaci.2008.11.019. Epub 2009 Jan 8. PMID 19135235